CLINICAL TRIAL: NCT02826720
Title: Is There a Relationship Between Hyperlipidemia and Periodontitis?
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MIHS-25
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Hyperlipidemia, Periodontal Disease
Keywords: HDL cholesterol; Hyperlipidemia; LDL cholesterol; Periodontal disease; Triglyceride
MeSH Terms: conditions — Hyperlipidemias; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- HP+: Subjects with plasma Triglyceride or Total cholesterol levels > 200 mg/dl and low density lipoprotein-cholesterol levels > 130 mg/dl were included in the hyperlipidemic group and having periodontitis which were further evaluated for clinical periodontal parameters as well as to define the effects of the patient's habits on plasma lipid levels.
  Interventions: Other: No intervention was applied
- HP-: Subjects with plasma Triglyceride or Total cholesterol levels > 200 mg/dl and low density lipoprotein-cholesterol levels > 130 mg/dl were included in the hyperlipidemic group and do not have periodontitis which were further evaluated for clinical periodontal parameters as well as to define the effects of the patient's habits on plasma lipid levels.
  Interventions: Other: No intervention was applied
- NP+: Subjects with plasma Triglyceride or Total cholesterol levels < 200 mg/dl and low density lipoprotein-cholesterol levels < 130 mg/dl were included in the normolipidemic group and having periodontitis which were further evaluated for clinical periodontal parameters as well as to define the effects of the patient's habits on plasma lipid levels.
  Interventions: Other: No intervention was applied
- NP-: Subjects with plasma Triglyceride or Total cholesterol levels < 200 mg/dl and low density lipoprotein-cholesterol levels < 130 mg/dl were included in the normolipidemic group and do not have periodontitis which were further evaluated for clinical periodontal parameters as well as to define the effects of the patient's habits on plasma lipid levels.
  Interventions: Other: No intervention was applied

INTERVENTIONS:
Other: No intervention was applied — No intervention was applied

SUMMARY:
The aim of present study is to investigate any relationship between hyperlipidemia and periodontal disease regarding the periodontal parameters and plasma lipid parameters, along with age, gender, brushing habit, body mass index, dietary habit, physical activity, alcohol consumption.

In this cross sectional study, a total of 160 individuals were divided into two groups based on their metabolic status: hyperlipidemic group (n=97) and normolipidemic group (n=63). Plaque index, gingival index, bleeding on probing (BOP), probing depth (PD), clinical attachment level (CAL) clinical parameters and community periodontal index of treatment needs (CPITN) scores were measured. Triglyceride (TG), total cholesterol (TC), low density lipoprotein-cholesterol (LDL-C) and high density lipoprotein-cholesterol (HDL-C) levels had been determined previously during individuals routine systemic examinations. Daily brushing habits and interdental cleaning together with dietary habits, alcohol consumption and physical activity levels were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having no periodontal treatment within previous 6 months,
* number of natural teeth ≥ 10,
* no history of cancer and systemic disease that affects lipid levels or periodontium,
* no history of medical treatment for hyperlipidemia, BMI< 30 kg/m2,
* no pregnancy,
* no history of systemic antibiotic treatment within previous 3 months,
* no smoking.

Exclusion Criteria:

* patients with history of systemic disease that affects lipid metabolism or periodontal disease
* history of medical treatment for hyperlipidemia
* pregnancy, lactation or hormone replacement therapy at the time of study
* use of any other drug known to affect lipid metabolism or periodontal disease
* systemic infection or any history of systemic antibiotic treatment in previous 3 months
* smokers as well as ex-smokers

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 240 subjects were examined among patients who attended to the Department of Periodontology, Marmara University or the Turkish Heart Foundation and had their plasma lipid values determined within the last 3 months. Out of 240, 160 subjects (57 male, 103 female, age range 35-65 years) eligible for this study were selected.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Triglyceride (TG) | day 0
  Subjects with plasma TG or TC levels > 200 mg/dl and LDL-C levels > 130 mg/dl were included in the hyperlipidemic group, while the normolipidemic group comprised of patients with plasma TG or TC levels below the aforementioned limits
Total cholesterol (TC) | day 0
  Subjects with plasma TG or TC levels > 200 mg/dl and LDL-C levels > 130 mg/dl were included in the hyperlipidemic group, while the normolipidemic group comprised of patients with plasma TG or TC levels below the aforementioned limits
Low density lipoprotein cholesterol (LDL-C) | day 0
  Subjects with plasma TG or TC levels > 200 mg/dl and LDL-C levels > 130 mg/dl were included in the hyperlipidemic group, while the normolipidemic group comprised of patients with plasma TG or TC levels below the aforementioned limits

SECONDARY OUTCOMES:
Plaque index | day 0
  The measurement of the state of oral hygiene based on recording dental plaque accumulation
Gingival index | day 0
  An assessment level of gingival health and inflammation
Bleeding on probing | day 0
  A sign of gingival inflammation were assessed on the buccal, lingual, mesial and distal sites of each tooth
Probing depth | day 0
  The distance from the gingival margin to bottom of the pocket with using 0.5 mm diameter periodontal probe at mesiobuccal, midbuccal, distobuccal, distolingual, midlingual and mesiolingual sites of each tooth
Clinical attachment level | day 0
  The distance between the cemento-enamel junction and bottom of the pocket
Community Periodontal Index of Treatment Needs score | day 0
  These scores are used to represent healthy periodontium, bleeding after probing, dental calculus detected by probing, 4-5 mm deep pockets and deep pockets ≥ 6 mm, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Gülin Tulu Katı, PhD, Principal Investigator — Periodontist in Private Practice., Istanbul, Turkey. (E-mail: gulintulu@gmail.com); Ülkü Noyan, Prof. Dr., Study Chair — Periodontist in Private Practice., Istanbul, Turkey. (E-mail: noyanulku@yahoo.com); Bahar Kuru, Prof. Dr., Study Chair — Department of Periodontology, Faculty of Dentistry, Yeditepe University, Istanbul, Turkey. (E-mail: baharkuru@gmail.com); Leyla Kuru, Prof. Dr., Study Director — Department of Periodontology, Faculty of Dentistry, Marmara University, Istanbul, Turkey. (E-mail: lkuru@marmara.edu.tr); Ömer Birkan Ağralı, PhD, Study Chair — Department of Periodontology, Faculty of Dentistry, Marmara University, Istanbul, Turkey. (omer.agrali@marmara.edu.tr); Hatice Selin Yıldırım, PhD, Study Chair — Department of Periodontology, Faculty of Dentistry, Marmara University, Istanbul, Turkey. (Email: yildirimselin@hotmail.com)